CLINICAL TRIAL: NCT02886767
Title: Effects of Father-Neonate Skin-to-Skin Contact on Attachment: A Randomised Controlled Trial
Brief Title: Effects of Father-Neonate Skin-to-Skin Contact on Attachment
Acronym: FNSSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Er-Mei Chen, Head Nurse and graduate student of NTUNHS, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGH-P101077
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Parent-Child Relations
Keywords: skin to skin contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- skin-to-skin contact (SSC) (Experimental): Experimental: a daily skin-to-skin contact (SSC) at least 15 minutes in length
  Interventions: Other: skin to skin contact
- Control: hospital routine care (No Intervention): As the hospital routine. Allow the father to visit the neonate, touching the neonate

INTERVENTIONS:
Other: skin to skin contact — The researchers facilitated initial SSC between intervention-group participants and their infants within 24 hours of birthing under conditions that did not adversely affect spontaneous mother-infant SSC nor interfere with the early initiation of breastfeeding. Because it is standard practice to discharge vaginal-birth mothers on the third postpartum day, this study implemented the intervention during the first three postpartum days for both vaginal and cesarean birth cases.
  Arms: skin-to-skin contact (SSC)

SUMMARY:
This study examines the effect of skin-to-skin contact between father and newborn on the father-neonate attachment relationship. By block randomization, participants were allocated to an experimental (n=41) or a control group (n=42).

DETAILED DESCRIPTION:
This study examines how skin-to-skin contact between father and newborn affects the attachment relationship. A randomized controlled trial was conducted at a regional teaching hospital and a maternity clinic in northern Taiwan. The study recruited 83 first-time fathers aged 20 years or older. By block randomization, participants were allocated to an experimental (n=41) or a control group (n=42). With the exception of skin-to-skin contact (SSC), participants from each group received the same standard care. Both groups also received an Early Childcare for Fathers nursing pamphlet. During the first three days postpartum, the intervention group members were provided a daily SSC intervention with their respective infants. Each intervention session lasted at least 15 minutes in length. The outcome measure was the Paternal Attachment Questionnaire (PAQ).

Four field experts of clinical obstetrics and pediatrics validated the developed father-neonate SSC intervention. A description of the intervention used in this study is as follows:

The researchers facilitated initial SSC between intervention-group participants and their infants within 24 hours of birthing under conditions that did not adversely affect spontaneous mother-infant SSC nor interfere with the early initiation of breastfeeding. Because it is standard practice to discharge vaginal-birth mothers on the third postpartum day, this study implemented the intervention during the first three postpartum days for both vaginal and cesarean birth cases.

Meanwhile, intervention-group participants were provided with the nursing pamphlet, Early Childcare for Fathers, and briefed on its contents at hospital admission. Upon delivery, each newborn infant received immediate SSC with the mother and was then provided neonatal nursing before being placed temporarily into an incubator for observation. After the infant was confirmed as being in a "quiet alert" state, defined as eyes open and bright, breathing normal, and sensitive and responsive to stimuli, a researcher led the father into the nursery, helped him hold his infant, and facilitated initial SSC. Immediately afterward, the researcher - in accordance with each participant's expressed preference - either withdrew from the room or observed the infant from an appropriate distance. Two further father-infant SSC sessions were held on day 2 and day 3, respectively, in either the nursery or maternity ward. The sessions took place in a secluded section of the nursery or ward about two hours after one of the daily feedings and only after the infant had been bathed, towel dried, and fitted with a diaper. The session space included a comfortable armchair, a footrest, a partition screen, a pillow, and a towel or blanket. The ambient temperature was held at a constant 25~27°C.

Prior to touching their infant, participants wore a loose-fitting, front-button shirt or hospital smock and washed their hands. They then sat in the provided armchair and exposed their chest. A pillow and footrest were also made available for use. After the researcher confirmed the safety of all preparations, participants were given their infant to hold. The infant was cradled on the participant's chest in a fetal position, with the head held upwards either vertically or at a 30~60° angle. The exposed back of the infant was then covered by a blanket or clothing. The participant supported the infant with his hands placed on the infant's shoulder and back. Next, he made eye contact with the infant. Touch and soft voice contact commenced only after the infant was appropriately relaxed, as indicated by relaxed eyebrows, forehead, and chin muscles; slightly curled hands; a comfortably curled body position; and calm smile.18 Previous studies found that infants feel most at ease within 15 minutes of SSC with their parents and that verbal and non-verbal communication typically commences within this time period as well.16, 20 Thus, the researchers defined the minimum duration of SSC sessions as 15 minutes, with sessions longer than this duration allowed to continue until either consciously ended by the father or interrupted by other infant-care priorities.

After receiving institutional review board (IRB) approval for this study in November 2012, a random allocation computer program generated a random stratified allocation table that was used to direct participant recruitment.23 Upon hospital admission, participants in both the intervention and control groups received the Early Childcare for Fathers nursing pamphlet in order to promote understanding of early infant care and complete the pretest PAQ instrument. Afterward, intervention-group participants were orally briefed on pamphlet contents and shown how to successfully perform father-infant SSC. These participants subsequently engaged in at least one >15-minute SSC session with their infant on each of the first three postpartum days. On the other hand, control-group participants received only standard nursing care after receiving the pamphlet. After the 3-day study period, all participants completed and submitted the demographic survey form and post-test PAQ.

ELIGIBILITY:
Inclusion Criteria:

* older than 20 years;
* be at the hospital daily until discharge;
* be a nonsmoker;
* not have an alcohol addiction or be diagnosed with a psychological disorder; and
* sign an informed consent agreement.

Exclusion Criteria:

* the neonate gestational age less than 37 weeks;
* the neonate vital signs unstable; and
* the neonate with congenital abnormalities or diseases.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Paternal Attachment measured by the Paternal Attachment Questionnaire (PAQ) | the first three postpartum days
  measured by the Paternal Attachment Questionnaire (PAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Huei Kao, PhD, Study Director — National Taipei University of Nursing and Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shorey S, He HG, Morelius E. Skin-to-skin contact by fathers and the impact on infant and paternal outcomes: an integrative review. Midwifery. 2016 Sep;40:207-17. doi: 10.1016/j.midw.2016.07.007. Epub 2016 Jul 5. PMID 27476026
- [Result] Cong X, Ludington-Hoe SM, Hussain N, Cusson RM, Walsh S, Vazquez V, Briere CE, Vittner D. Parental oxytocin responses during skin-to-skin contact in pre-term infants. Early Hum Dev. 2015 Jul;91(7):401-6. doi: 10.1016/j.earlhumdev.2015.04.012. Epub 2015 May 16. PMID 25988992
- [Result] Nimbalkar A, Patel D, Sethi A, Nimbalkar S. Effect of skin to skin care to neonates on pulse rate, respiratory rate SPO2 and blood pressure in mothers. Indian J Physiol Pharmacol. 2014 Apr-Jun;58(2):174-7. PMID 25509971
- [Result] Moore ER, Anderson GC, Bergman N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003519. doi: 10.1002/14651858.CD003519.pub2. PMID 17636727
- [Result] Cho ES, Kim SJ, Kwon MS, Cho H, Kim EH, Jun EM, Lee S. The Effects of Kangaroo Care in the Neonatal Intensive Care Unit on the Physiological Functions of Preterm Infants, Maternal-Infant Attachment, and Maternal Stress. J Pediatr Nurs. 2016 Jul-Aug;31(4):430-8. doi: 10.1016/j.pedn.2016.02.007. Epub 2016 Mar 11. PMID 26975461
- [Result] Stevens J, Schmied V, Burns E, Dahlen H. Immediate or early skin-to-skin contact after a Caesarean section: a review of the literature. Matern Child Nutr. 2014 Oct;10(4):456-73. doi: 10.1111/mcn.12128. Epub 2014 Apr 10. PMID 24720501
- [Result] Conde-Agudelo A, Belizan JM, Diaz-Rossello J. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD002771. doi: 10.1002/14651858.CD002771.pub2. PMID 21412879
- [Result] Lee SB, Shin HS. [Effects of Kangaroo Care on anxiety, maternal role confidence, and maternal infant attachment of mothers who delivered preterm infants]. Taehan Kanho Hakhoe Chi. 2007 Oct;37(6):949-56. doi: 10.4040/jkan.2007.37.6.949. Korean. PMID 17992067
- [Result] Wang YH, Kuo HH. [The nursing experience in helping an unmarried adolescence girl to care for her premature infant]. Hu Li Za Zhi. 2006 Oct;53(5):76-83. Chinese. PMID 17004211
- [Derived] Chen EM, Gau ML, Liu CY, Lee TY. Effects of Father-Neonate Skin-to-Skin Contact on Attachment: A Randomized Controlled Trial. Nurs Res Pract. 2017;2017:8612024. doi: 10.1155/2017/8612024. Epub 2017 Jan 17. PMID 28194281